CLINICAL TRIAL: NCT00502996
Title: Multicenter Non-Comparative Expanded Access Program of to Assess Safety of Rituximab (Mab Anti Cd-20) in Patients With Rheumatoid Arthritis (Ser)
Brief Title: A Non-Comparative Study to Assess the Safety of MabThera (Rituximab) in Patients With Rheumatoid Arthritis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19385
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Results first posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Rituximab

ARMS (1):
- Rituximab (Experimental): Eligible participants receiving Rituximab (MabThera/Rituxan) 1 gram/dose (g/dose) intravenously (IV) on Day 1 and Day 15 followed by previous pre-medication (methylprednisolone 100 mg IV, antihistamine and antipyretic) and concomitant treatment of Methotrexate at least 15 mg per oris (PO) weekly were observed during the study period of 24 weeks. After treatment completion, participants were followed-up for safety up to 24 weeks.
  Interventions: Drug: Methotrexate; Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: Methotrexate — >=15 mg po/week
Drug: rituximab [MabThera/Rituxan] — 1g iv on days 1 and 15

SUMMARY:
This single arm study will assess the safety of MabThera plus methotrexate in patients with rheumatoid arthritis who have had a lack of response to 1-5 DMARDs or biological agents. Patients will receive MabThera (1g i.v.) on days 1 and 15, concomitantly with methotrexate >=15mg p.o./week. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* rheumatoid arthritis >=6 months;
* lack of response to 1-5 DMARDs or biological agents;
* rheumatoid factor positive.

Exclusion Criteria:

* other chronic inflammatory articular disease or systemic rheumatic disease;
* joint or bone surgery during 8 weeks prior to randomization;
* previous treatment with any cell-depleting therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - San Miguel de Tucumán
- Brazil (15):
  - Belém
  - Brasília
  - Campinas
  - Curitiba
  - Florianópolis
  - Fortaleza
  - Goiânia
  - Nova Lima
  - Porto Alegre
  - Recife
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - São Paulo
  - Vitória
- Santiago, Chile
- Colombia (2):
  - Barranquilla
  - Bogotá
- Ecuador (3):
  - Cuenca
  - Guayaquil
  - Quito
- San Salvador, El Salvador
- Mexico (2):
  - Mexico City
  - San Luis Potosí City
- Peru (3):
  - Jesus Maria
  - Lima
  - San Isidro
- Montevideo, Uruguay
- Venezuela (2):
  - Barquisimeto
  - Caracas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 246 participants were enrolled in study conducted from 20 February 2006 to 05 December 2008 across 56 study centers in 10 Latin American countries.
Pre-assignment Details: Out of 246 participants, fourteen did not receive study drug and were not included in analysis population.
Groups:
- Rituximab: Eligible participants receiving Rituximab (MabThera/Rituxan) 1 gram/dose (g/dose) intravenously (IV) on Day 1 and Day 15 followed by previous pre-medication (methylprednisolone 100 milligram (mg) IV, antihistamine and antipyretic) and concomitant treatment of Methotrexate at least 15 mg per oris (PO) weekly were observed during the study period of 24 weeks. After treatment completion, participants were followed-up for safety up to 24 weeks.
Period: Overall Study
Arm/Group | Rituximab
Started | 232
Completed | 188
Not Completed | 44
Not completed — Lost to Follow-up | 9
Not completed — Protocol Violation | 2
Not completed — Treatment failure | 25
Not completed — Withdrawal Informed Consent | 6
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: The safety population included all eligible participants who received one treatment dose of rituximab and have completed the follow up period (Week 48) regardless of whether withdrawn or not from the study.
Groups:
- Rituximab: Eligible participants receiving Rituximab 1 g/dose IV on Day 1 and Day 15 followed by previous pre-medication (methylprednisolone 100 mg IV, antihistamine and antipyretic) and concomitant treatment of Methotrexate at least 15 mg PO weekly were observed during the study period of 24 weeks. After treatment completion, participants were followed-up for safety up to 24 weeks.
Arm/Group | Rituximab
Number analyzed (Participants) | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event, Any Serious Adverse Event, and Death
Description: An Adverse event (AE) was considered any unfavorable medical event in a participant of clinical research who received the study drug and that not necessarily had a causal relationship with this treatment. An AE could, therefore, being any unfavorable sign and non-intentional, symptom or disease temporarily related with the use of a medicinal product, considered or not related to the medicinal product. Pre-existing conditions that worsened during the study were reported as AEs. A serious adverse event (SAE) is any experience that suggested a significant risk, contraindication, caution, and at any dose fulfills at least one of the following criteria: adverse event considered as fatal (resulting in death), life threatening, defect of birth/congenital abnormality, required hospitalization or extension of hospital length of stay, significant medical intervention, resulted in significant disability/impairment.
Time Frame: Up to Week 48
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 232
participants
  Any AE | 189
  Any SAE | 12
  Death | 0

2. Primary Outcome: Number of Participants With AEs According to Degree of Intensity
Description: An AE is any unfavorable sign and non-intentional, symptom or disease temporarily related with the use of a medicinal product, considered or not related to the medicinal product. Pre-existing conditions that worsened during the study were reported as AEs. The Intensity of AEs was classified as Grade 1, Grade 2, Grade 3 and Grade 4. Grade 1: Discomfort was noticed, but the normal daily activity was not interrupted. Grade 2: Discomfort was enough to reduce the normal daily activity. Grade 3: There was disability for work or develop normal daily activities. Grade 4: It represented an immediate threat to life (these events were reported as SAEs).
Time Frame: Up to Week 48
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 232
participants
  Grade 1 AEs | 170
  Grade 2 AEs | 102
  Grade 3 AEs | 30
  Grade 4 AEs | 12

3. Primary Outcome: Number of Participants With AEs Leading to Discontinuation and Any Drug Related AEs and SAEs
Description: An AE is any unfavorable sign and non-intentional, symptom or disease temporarily related with the use of a medicinal product, considered or not related to the medicinal product. Pre-existing conditions that worsened during the study were reported as AEs. A SAE is any experience that suggested a significant risk, contraindication, caution, and at any dose, fulfills, at least, one of the following criteria: adverse event considered as fatal (resulting in death), life threatening, defect of birth/congenital abnormality, required hospitalization or extension of hospital length of stay, significant medical intervention, resulted in significant disability/impairment. Relationship between AEs and medication under investigation was evaluated through the classification "Yes" and "No". A relationship classified as "Yes" implied a significant causal relationship with the medication under investigation which was evaluated based on enough evidences, facts or arguments.
Time Frame: Up to Week 48
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 232
participants
  Any drug related AE | 97
  Any drug related SAE | 0
  Any AE leading to discontinuation | 2

4. Primary Outcome: Number of Participants With AEs of Special Interest During the Study
Description: Adverse event of special interest during the study treatment and follow up period included infections. The participants with AEs of special interest were reported at Screening, End of treatment (EOT), and End of Follow-up (EOFU) visit.
Time Frame: Screening (Days -28 to 0), EOT (Week 24), and EOFU (Week 48)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 232
participants
  Screening | 5
  EOT | 12
  EOFU | 12

5. Secondary Outcome: Mean Values of Hematology Parameters at Screening and EOT Visit (Hemoglobin and Mean Corpuscular Hemoglobin Concentration)
Description: The values of hemoglobin (Hb) and mean corpuscular hemoglobin concentration (MCHC) for each participant were estimated at Screening and at EOT visit.
Time Frame: Screening (Days -28 to 0) and EOT (Week 24)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/deciliter (dL)
Arm/Group | Rituximab
Number analyzed (Participants) | 191
g/deciliter (dL)
  Hb, Screening | 12.4 (1.9)
  Hb, EOT | 12.8 (1.6)
  MCHC, Screening | 30.0 (3.6)
  MCHC, EOT | 30.9 (2.7)

6. Secondary Outcome: Mean Values of Hematology Parameters at Screening and EOT Visit (Hematocrit, Neutrophils, Lymphocytes, Monocytes, Eosinophils, and Basophils)
Description: The hematology parameters (hematocrit, neutrophils, lymphocytes, monocytes, eosinophils, and basophils) for each participant were estimated at Screening and at EOT.
Time Frame: Screening (Days -28 to 0) and EOT (Week 24)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Rituximab
Number analyzed (Participants) | 191
percentage of cells
  Hematocrit, Screening | 37.8 (4.2)
  Hematocrit, EOT | 38.9 (4.3)
  Neutrophils, Screening | 67.8 (9.4)
  Neutrophils, EOT | 65.1 (9.9)
  Lymphocytes, Screening | 24.0 (7.7)
  Lymphocytes, EOT | 25.6 (8.7)
  Monocytes, Screening | 4.3 (3.1)
  Monocytes, EOT | 5.4 (3.6)
  Eosinophils, Screening | 1.9 (2.0)
  Eosinophils, EOT | 2.5 (2.0)
  Basophils, Screening | 0.2 (0.3)
  Basophils, EOT | 0.3 (0.4)

7. Secondary Outcome: Mean Values of Hematology Parameter at Screening and EOT Visit (Mean Corpuscular Volume)
Description: Mean corpuscular volume (MCV) is the average volume of red cells. The mean MCV concentration for each participant was estimated at Screening and EOT.
Time Frame: Screening (Days -28 to 0) and EOT (Week 24)
Population: The analysis was performed on safety population. Eligible participants who received one treatment dose of Rituximab, have completed the follow-up period, Visit 11, and end of follow-up period in safety conditions and also who had been withdrawn or not from the study were included in the safety population.
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Rituximab
Number analyzed (Participants) | 191
femtoliters
  MCV, Screening | 85.8 (8.5)
  MCV, EOT | 87.7 (7.0)

8. Secondary Outcome: Mean Values of Hematology Parameter at Screening and EOT Visit (Erythrocytes)
Description: The mean erythrocyte concentration for each participant was estimated at Screening and at EOT.
Time Frame: Screening (Days -28 to 0) and EOT (Week 24)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Rituximab
Number analyzed (Participants) | 191
10^12 cells/liter
  Erythrocytes, Screening | 4.5 (1.2)
  Erythrocytes, EOT | 4.4 (0.5)

9. Secondary Outcome: Mean Values of Hematology Parameters at Screening and EOT Visit (Leucocytes and Platelets)
Description: The mean leucocytes and platelets concentration for each participant was estimated at Screening, at EOT visit.
Time Frame: Screening (Days -28 to 0) and EOT (Week 24)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Rituximab
Number analyzed (Participants) | 191
10^9 cells/liter
  Leucocytes, Screening | 8.6 (2.6)
  Leucocytes, EOT | 7.7 (2.3)
  Platelets, Screening | 351.6 (112.5)
  Platelets, EOT | 310.6 (97.1)

10. Secondary Outcome: Mean Values of Biochemistry Parameters at Screening and Visit 8 (Albumin and Glucose)
Description: The mean albumin and glucose concentration for each participant was estimated at Screening and at EOT visit.
Time Frame: Screening (Days -28 to 0) and EOT (Week 24)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Rituximab
Number analyzed (Participants) | 191
g/dL
  Albumin, Screening | 3.9 (0.5)
  Albumin, EOT | 4.1 (0.4)
  Glucose, Screening | 86.1 (12.3)
  Glucose, EOT | 88.1 (26.5)

11. Secondary Outcome: Mean Values of Cholesterol, Uric Acid, Urea, Creatinine, Calcium, Total Bilirubin and Serum Total Proteins at Screening and EOT Visit.
Description: The mean concentration of cholesterol, uric acid, urea, creatinine, calcium, total bilirubin and serum total proteins (STP) for each participant was estimated at Screening and at EOT visit.
Time Frame: Screening (Days -28 to 0) and EOT (Week 24)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rituximab
Number analyzed (Participants) | 191
mg/dL
  Cholesterol, Screening | 187.9 (42.2)
  Cholesterol, EOT | 196.6 (42.7)
  Uric acid, Screening | 4.0 (1.2)
  Uric acid, EOT | 4.0 (1.1)
  Urea, Screening | 29.3 (10.0)
  Urea, EOT | 30.2 (11.0)
  Creatinine, Screening | 0.7 (0.2)
  Creatinine, EOT | 0.7 (0.2)
  Calcium, Screening | 9.0 (1.3)
  Calcium, EOT | 9.0 (1.0)
  Total Bilirubin, Screening | 0.7 (1.1)
  Total Bilirubin, EOT | 0.7 (1.1)
  STP, Screening | 7.3 (0.6)
  STP, EOT | 7.1 (0.6)

12. Secondary Outcome: Mean Values of Potassium, Chlorine, Sodium, and Phosphorus at Screening and EOT Visit
Description: The mean concentration of potassium, chlorine, sodium and phosphorus for each participant was estimated at Screening and at EOT.
Time Frame: Screening (Days -28 to 0) and EOT (Week 24)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Rituximab
Number analyzed (Participants) | 191
millimoles per liter
  Sodium, Screening | 140.1 (3.3)
  Sodium, EOT | 140.4 (3.3)
  Potassium, Screening | 4.2 (0.4)
  Potassium, EOT | 4.2 (0.4)
  Chlorine, Screening | 103.1 (4.2)
  Chlorine, EOT | 103.3 (4.2)
  Phosphorus, Screening | 3.7 (0.6)
  Phosphorus, EOT | 3.8 (0.7)

13. Secondary Outcome: Mean Values of Aspartate Transaminase, Alanine Transaminase, Alkaline Phosphatase, and Lactic Dehydrogenase at Screening and EOT Visit
Description: The mean aspartate transaminase (AST) and alanine transaminase (ALT), Alkaline phosphatase (AP), and Lactic dehydrogenase (LDH) concentration for each participant was estimated at Screening and at EOT visit.
Time Frame: Screening (Days -28 to 0) and EOT (Week 24)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: International units/liter
Arm/Group | Rituximab
Number analyzed (Participants) | 191
International units/liter
  AST, Screening | 21.6 (9.7)
  AST, EOT | 22.0 (9.5)
  ALT, Screening | 24.1 (14.9)
  ALT, EOT | 25.9 (14.9)
  AP, Screening | 137.7 (71.6)
  AP, EOT | 138.2 (81.7)
  LDH, Screening | 311.0 (149.1)
  LDH, EOT | 300.5 (125.4)

14. Secondary Outcome: Mean Duration of Morning Joint Stiffness
Description: The efficacy of rituximab was assessed by evaluating mean duration of morning joint stiffness.
Time Frame: Screening ((Days -28 to 0), EOT (Week 24), and EOFU (Week 48)
Population: All eligible participants who received one treatment dose of rituximab were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rituximab
Number analyzed (Participants) | 232
Minutes
  Screening | 120.1 (96.3)
  EOT | 16.0 (36.5)
  EOFU | 19.9 (42.4)

15. Secondary Outcome: Mean Value of Painful Joints
Description: The efficacy of rituximab was assessed by evaluating painful joints.
Time Frame: Screening (Days -28 to 0), EOT (Week 24), and EOFU (Week 48)
Population: All eligible participants who received one treatment dose of rituximab were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: number of painful joints
Arm/Group | Rituximab
Number analyzed (Participants) | 232
number of painful joints
  Painful joints, Screening | 17.5 (8.6)
  Painful joints, EOT | 3.8 (4.9)
  Painful joints, EOFU | 4.4 (5.7)

16. Secondary Outcome: Number of Participants With American College of Rheumatology (20, 50, and 70) Criteria
Description: American College of Rheumatology (ACR) criteria improvement consisting of 20%, 50%, and 70% (ACR20, ACR50, and ACR70, respectively) reduction in tender joints and swollen joints, as well as for three of the additional five ACR core set variables: patient's assessment of pain using a Visual Analog Scale (VAS) with left end of the line 0=no pain to right end of the line 100=unbearable pain); patient's global assessment of disease activity and physician's global assessment of disease activity using a VAS (0=no disease activity to 100=maximum disease activity); health assessment questionnaire (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant; C-reactive protein and globular sedimentation velocity.
Time Frame: Week 1, Week 12, and Week 24
Population: All eligible participants who received one treatment dose of rituximab were considered for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 232
participants
  ACR 20, Week 1 | 1
  ACR 20, Week 12 | 84
  ACR 20, Week 24 | 88
  ACR 50, Week 1 | 0
  ACR 50, Week 12 | 50
  ACR 50, Week 24 | 62
  ACR 70, Week 1 | 0
  ACR 70, Week 12 | 33
  ACR 70, Week 24 | 42

17. Secondary Outcome: Mean Value of Quality of Life (Health Assessment Questionnaire - Disease Index)
Description: Health Assessment Questionnaire - Disease Index (HAQ-DI) indicates how the disease affected participant's activities of daily life. It consisted of 20 questions in 8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities) rated on a 4-point scale, 0=without any difficulty to 3=unable to do. Sum of scores was divided by number of domains with a score for a total possible score of 0 (best/no difficulties to perform activities) to 3 (worst/ unable to perform activities at all).
Time Frame: Screening (Days -28 to 0), Week 1, Week 12, and Week 24
Population: All eligible participants who received one treatment dose of rituximab were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Rituximab
Number analyzed (Participants) | 106
Scores on scale
  Screening; n = 106 | 2.6 (1.3)
  Week 1; n = 114 | 2.5 (1.4)
  Week 12; n = 107 | 1.25 (1.0)
  Week 24; n = 105 | 1.0 (1.0)

18. Secondary Outcome: Mean Values of C Reactive Protein
Description: C Reactive Protein (CRP) is a component of ACR. CRP is a marker of inflammation.
Time Frame: Screening ((Days -28 to 0), EOT (Week 24), and EOFU (Week 48)
Population: All eligible participants who received one treatment dose of rituximab were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams per liter
Arm/Group | Rituximab
Number analyzed (Participants) | 232
milligrams per liter
  Screening | 28.0 (45.3)
  Week 1 | 27.6 (56.1)
  Week 12 | 13.6 (25.0)
  Week 24 | 15.3 (45.2)

19. Secondary Outcome: Mean Values of Globular Sedimentation Velocity
Description: Globular sedimentation velocity is a component of ACR.
Time Frame: Screening ((Days -28 to 0), Week 1, Week 12, and Week 24
Population: All eligible participants who received one treatment dose of rituximab were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeters per hour
Arm/Group | Rituximab
Number analyzed (Participants) | 232
millimeters per hour
  Screening | 43.7 (22.8)
  Week 1 | 41.1 (23.0)
  Week 12 | 26.8 (17.8)
  Week 24 | 24.6 (19.0)

20. Secondary Outcome: Mean Values of Pain and Activity Based on Visual Analogue Scale
Description: Pain assessment was assessed by using a VAS (0=no pain to 100=unbearable pain). Disease activity was also evaluated by participants and investigators by using a VAS (0=no disease activity to 100=maximum disease activity).
Time Frame: Screening ((Days -28 to 0), Week 1, Week 12, and Week 24
Population: All eligible participants who received one treatment dose of rituximab were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Rituximab
Number analyzed (Participants) | 232
Scores on scale
  Pain, Screening | 6.9 (1.9)
  Pain, Week 1 | 6.9 (1.9)
  Pain, Week 12 | 3.6 (2.4)
  Pain, Week 24 | 3.0 (2.2)
  Activity (participant), Screening | 6.6 (2.3)
  Activity (participant), Week 1 | 5.9 (2.5)
  Activity (participant), Week 12 | 4.7 (2.8)
  Activity (participant), Week 24 | 3.9 (2.7)
  Activity (investigator), Screening | 6.4 (2.0)
  Activity (investigator), Week 1 | 6.3 (2.1)
  Activity (investigator), Week 12 | 3.9 (3.9)
  Activity (investigator), Week 24 | 3.0 (2.5)

21. Secondary Outcome: Mean Value of Inflamed Joints
Description: The efficacy of rituximab was assessed by evaluating inflamed joints.
Time Frame: Screening (Days -28 to 0), EOT (Week 24), and EOFU (Week 48)
Population: All eligible participants who received one treatment dose of rituximab were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: number of inflamed joints
Arm/Group | Rituximab
Number analyzed (Participants) | 232
number of inflamed joints
  Inflamed joints, Screening | 17.5 (8.6)
  Inflamed joints, EOT | 3.8 (4.9)
  Inflamed joints, EOFU | 4.4 (5.7)

ADVERSE EVENTS:
Time Frame: Up to Week 48
Description: Safety population was used for collecting data on adverse events. The safety population included all eligible participants who received one treatment dose of rituximab and, have completed the follow up period (Week 48) regardless of whether withdrawn or not from the study.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 12/232
Other Adverse Events (participants affected / at risk) | 189/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=232)
Abdominal distension (Gastrointestinal disorders) | 1
Acute gastroenteritis (Gastrointestinal disorders) | 1
Ovarian neoplasm NOS (Reproductive system and breast disorders) | 1
Uterine myoma (Reproductive system and breast disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Tubo-ovarian abscess (Infections and infestations) | 1
Arthritis aggravated (Musculoskeletal and connective tissue disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Acute kidney failure (Renal and urinary disorders) | 1
Baker's cyst excision (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=232)
Nausea (Gastrointestinal disorders) | 22
Diarrhea (Gastrointestinal disorders) | 16
Dyspepsia (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 9
Gastritis (Gastrointestinal disorders) | 9
Pyrosis (Gastrointestinal disorders) | 6
Epigastralgia (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 4
Epigastric burning (Gastrointestinal disorders) | 4
Colitis (Gastrointestinal disorders) | 3
Dry throat (Gastrointestinal disorders) | 3
Urinary tract infection (Infections and infestations) | 23
Upper respiratory tract infection viral NOS (Infections and infestations) | 14
Pharyngitis (Infections and infestations) | 9
Bronchitis (Infections and infestations) | 5
Tonsillitis (Infections and infestations) | 4
Tooth infection (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 3
Cold (Respiratory, thoracic and mediastinal disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 7
Lower respiratory tract infection NOS (Respiratory, thoracic and mediastinal disorders) | 6
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 6
Dry cough (Respiratory, thoracic and mediastinal disorders) | 3
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Headache (Nervous system disorders) | 40
Dizziness (Nervous system disorders) | 17
Vertigo (Nervous system disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 7
Accelerated hair loss (Skin and subcutaneous tissue disorders) | 6
Pruritus NOS (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 4
Skin rash (Skin and subcutaneous tissue disorders) | 4
Skin ulcer NOS (Skin and subcutaneous tissue disorders) | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Itching (Skin and subcutaneous tissue disorders) | 3
Low back pain (Musculoskeletal and connective tissue disorders) | 8
Arthritis aggravated (Musculoskeletal and connective tissue disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Lumbago (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Shivers (General disorders) | 9
Disease progression (General disorders) | 6
Hyperthermia (General disorders) | 6
Fatigue (General disorders) | 3
Conjunctivitis (Eye disorders) | 6
Xerophthalmia (Eye disorders) | 4
Somnolence (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 5
Rheumatoid arthritis aggravated (Immune system disorders) | 5
Allergic conditions (Immune system disorders) | 3
Allergic rhinitis (Immune system disorders) | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3
Osteoporosis (Metabolism and nutrition disorders) | 3
Hypertension arterial (Vascular disorders) | 12
Dyspnea (Cardiac disorders) | 6
Arrhythmia (Cardiac disorders) | 3
Hematuria (Renal and urinary disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.